CLINICAL TRIAL: NCT03902236
Title: Evaluation of Reaction Time and Postural Control in Individuals With Cystic Fibrosis and Bronchiectasis
Brief Title: Reaction Time and Postural Control in Individuals With Cystic Fibrosis and Bronchiectasis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Jan Dik, Master of Science student, Hacettepe University
Other Study IDs: cfreactiontime
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Cystic Fibrosis; Bronchiectasis
Keywords: postural control; reaction time; cystic fibrosis; Bronchiectasis
MeSH Terms: conditions — Cystic Fibrosis; Bronchiectasis | interventions — Reaction Time; Postural Balance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cystic fibrosis group: Children diagnosed with cystic fibrosis more than 6 years old Stable medical condition Those who have not participated in a planned training program in the last 3 months
  Interventions: Other: Reaction Time and Postural Control; Other: Muscle oxygenation; Other: Exercise capacity; Other: Balance
- Bronchiectasis group: Children diagnosed with bronchiectasis more than 6 years old Stable medical condition Those who have not participated in a planned training program in the last 3 months
  Interventions: Other: Reaction Time and Postural Control; Other: Muscle oxygenation; Other: Exercise capacity; Other: Balance
- Healthy group: Healthy children more than 6 years old Stable medical condition Those who have not participated in a planned training program in the last 3 months
  Interventions: Other: Reaction Time and Postural Control; Other: Muscle oxygenation; Other: Exercise capacity; Other: Balance

INTERVENTIONS:
Other: Reaction Time and Postural Control — Reaction Time and Postural Control: With ''Fitlight TrainerTM'', 6 light emitting diode (LED) lights placed at certain points on the wall are randomly lit and expected to deactivate them as fast as possible. In the protocol, the leds will be placed according to the physical structure of the person, and the scores of 29 LED's will be kept in seconds. The scores will be compared cystic fibrosis, bronchiectasis and healthy groups.
Other: Muscle oxygenation — Muscle oxygenation will be assessed with wearable lactate threshold predicting device in cystic fibrosis, bronchiectasis and healthy groups.
Other: Exercise capacity — Exercise capacity will be assessed with incremental shuttle walk test in cystic fibrosis, bronchiectasis and healthy groups.The patient is required to walk around two cones set 9 metres apart (so the final track is 10 metres) in time to a set of auditory beeps played on a CD. Initially, the walking speed is very slow, but each minute the required walking speed progressively increases.The patient walks for as long as they can until they are either too breathless or can no longer keep up with the beeps, at which time the test ends The number of shuttles is recorded. Each shuttle represents a distance of ten metres
Other: Balance — Balance will be assessed with functional reach test in cystic fibrosis, bronchiectasis and healthy groups Functional Reach measures the maximum distance a person can reach forward, the distance of the person standing at the edge of the wall with a 90-degree shoulder flexion and the maximum distance to the front of the thumb will be noted.

SUMMARY:
The aim of this study is to evaluate the reaction time and postural control and to investigate the relationship between reaction time, exercise capacity, muscle oxygenation and balance in children with cystic fibrosis (CF) and non-CF bronchiectasis. 40 patients including 20 CF patients and 20 non-CF bronchiectasis and 20 healthy individuals will be included in this study. Demographic and physical characteristics' will be recorded. Lung function testing will be performed. Balance will be assessed using functional reach test, exercise capacity was measured using the incremental shuttle walking test and reaction time will be assessed using ''Fitlight TrainerTM''. Heart rate, respiratory rate, oxygen saturation, muscle oxygenation, dyspnea and fatigue perception will be measured before and after exercise test and reaction time measurement.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with bronchiectasis and cystic fibrosis at 6-18 years old age for the bronchiectasis and cystic fibrosis groups respectively
* Healthy children at 6-18 years old age for the healthy group.
* Stable medical condition (free from the acute exacerbation)
* Children who have not participated in the planned exercise training program in the last 3 months
* Compliance with the tests

Exclusion Criteria:

* Children who have a physical problems that limit the application of the tests
* Acute infection or unstable medical status

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children diagnosed with cystic fibrosis and bronchiectasis is referred from Hacettepe University, Pediatric Chest Diseases Department to Hacettepe University Department of Physiotheraphy and Rehabilitation will be included in this study. And also, healthy children at 6-18 years olds who are relatives of patients admitted to the our department will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-10-07 (Estimated); Study Completion 2019-11-04 (Estimated)

PRIMARY OUTCOMES:
Reaction Time and Postural Control | 8 minutes
  Reaction Time and Postural Control: With bunlar Fitlight TrainerTM muş, 6 led lights placed at certain points on the wall are randomly lit and expected to extinguish them as fast as possible. In the protocol, the leds will be placed according to the physical structure of the person, and the scores of 29 LEDs will be kept in seconds. The scores will be compared cystic fibrosis, bronciechtasis and healthy groups.
Muscle oxygenation | 40 minutes (during the incremental shuttle walk test+reaction and postural control protocol)
  Muscle oxygenation will be assessed with wearable lactate threshold predicting device in cystic fibrosis, bronciechtasis and healthy groups.
Exercise capacity | 20 minutes
  Exercise capacity will be assessed with incremental shuttle walk test in cystic fibrosis, bronciechtasis and healthy groups.The patient is required to walk around two cones set 9 metres apart (so the final track is 10 metres) in time to a set of auditory beeps played on a CD. Initially, the walking speed is very slow, but each minute the required walking speed progressively increases.The patient walks for as long as they can until they are either too breathless or can no longer keep up with the beeps, at which time the test ends The number of shuttles is recorded. Each shuttle represents a distance of ten metres
Balance | 5 minutes
  Balance will be assessed with functional reach test in cystic fibrosis, bronciechtasis and healthy groups Functional Reach measures the maximum distance a person can reach forward, the distance of the person standing at the edge of the wall with a 90-degree shoulder flexion and the maximum distance to the front of the thumb will be noted.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borges NR, Driller MW. Wearable Lactate Threshold Predicting Device is Valid and Reliable in Runners. J Strength Cond Res. 2016 Aug;30(8):2212-8. doi: 10.1519/JSC.0000000000001307. PMID 27457915
- [Background] Klein M, Gauggel S, Sachs G, Pohl W. Impact of chronic obstructive pulmonary disease (COPD) on attention functions. Respir Med. 2010 Jan;104(1):52-60. doi: 10.1016/j.rmed.2009.08.008. Epub 2009 Sep 11. PMID 19748260